CLINICAL TRIAL: NCT01613157
Title: Predictors of Antiretroviral Pharmacokinetics in HIV-infected Women With Virologic Suppression
Status: Completed | Type: Observational
Sponsor: Canadian Immunodeficiency Research Collaborative (Other)
Responsible Party: Sponsor
Other Study IDs: CIHR-PK1
Record Dates: First submitted 2009-11-05; First posted 2012-06-07 (Estimated); Last update posted 2012-06-07 (Estimated); Status verified 2012-06

CONDITIONS: Human Immunodeficiency Virus
Keywords: pharmacokinetics; HIV infected women
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
The investigators would like to carry out this study to measure drug levels in HIV-infected women that are taking anti-HIV medications. This study will determine the predictors of high drug levels and will assess the association of drug levels and adverse events in women.

DETAILED DESCRIPTION:
There have been tremendous advances in the treatment of HIV by combining 3 to 4 of the 20 anti-HIV medications available. Despite these advances, there remain several important complications related to the treatment, most importantly adverse events like nausea, diarrhea, liver toxicity and lipodystrophy (fat wasting or accumulation). Some studies have found that drug levels are higher in women and that these higher drug levels are associated with the increased toxicity in women. The reasons for the higher drug levels remain unclear. It is unknown whether these relate to hormonal influences, drug metabolism, adherence, fat distribution, body size or other factors. For this reason, we would like to carry out this study to measure drug levels in HIV-infected women that are taking anti-HIV medications. This study will determine the predictors of high drug levels and will assess the association of drug levels and adverse events in women.

ELIGIBILITY:
Inclusion Criteria:

* Are HIV infected
* Are 18 years old or older
* A biologic woman
* Are taking their first combination Anti-retroviral regimen that includes a Protease Inhibitor or a Non-Nucleoside Reverse Transcriptase Inhibitor for the past three months with no changes in any part of the combination in that period
* Are taking either a Protease Inhibitor or an Non-Nucleoside Reverse Transcriptase Inhibitor but not both
* If taking a Protease Inhibitor, must be taking only one Protease Inhibitor excluding low dose ritonavir used as boosting
* Have a viral load < 50 copies/mL on two occasions at least 1 month apart including a value at least three months before the baseline visit
* Have signed and dated a full informed consent

Exclusion Criteria:

* Have difficulty participating in a trial due to non-adherence or substance abuse
* Pregnant or breast-feeding
* Have malignancy receiving systemic chemotherapy
* Have end-stage organ disease
* Have another significant non-HIV underlying disease that might impinge upon disease progression or death

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HIV positive patients
Sampling Method: Non-Probability Sample
Enrollment: 88 (Actual)
Dates: Start 2006-01; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mona Loutfy, MD, Principal Investigator — Sunnybrook and Women's College Health Science Centre
Locations (1):
- Maple Leaf Medical Clinic, Toronto, Ontario, Canada